CLINICAL TRIAL: NCT00979472
Title: Comparison of the Effect of Flexible Dosage of Solifenacin Succinate Between Patients Who Have Frequent Micturition With and Without Urgency
Brief Title: Solifenacin Flexible Dosing Study in Frequent Micturition Patients With and Without Urgency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Principal Investigator, Myung-Soo Choo, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VC-2009-0014
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Urinary Bladder, Overactive; Overactive Bladder
Keywords: Solifenacin; Overactive bladder; Micturition; Urinary urgency; Vesicare
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with urgency (Experimental)
  Interventions: Drug: Solifenacin
- without urgency (Experimental)
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — oral
  Other Names: YM905; Vesicare

SUMMARY:
The purpose of the study is to compare the effect of solifenacin succinate between frequent micturition patients with urgency and those without urgency.

ELIGIBILITY:
Inclusion Criteria:

* For the without-urgency group:

  * urinary frequency ≥ 8 micturitions per 24 hours no urgency on voiding diary (1 or 2 on a 5 urgency scale)
* For the with-urgency group:

  * urinary frequency ≥ 8 micturitions per 24 hours symptoms of urinary urgency≥ 2/day on the voiding diary (3 to 5 on a 5 urgency scale)
* Symptoms lasting for more than 3 months

Exclusion Criteria:

* Clinically significant stress incontinence as determined by the investigator; for female patients, clinically significant stress incontinence confirmed by a cough provocation test
* Total daily urine volume of > 3000 mL as verified on the micturition diary before randomization
* Significant hepatic or renal disease, defined as having twice the upper limit of the reference ranges for serum concentrations of aspartate aminotra
* Any condition that is a contraindication for anticholinergic treatment, including uncontrolled narrow-angled glaucoma, urinary retention or gastric retention
* Symptomatic acute urinary tract infection (UTI) during the run-in period
* Recurrent UTIs defined as having been treated for symptomatic UTIs > 4 times in the last year
* Diagnosed or suspected of interstitial cystitis
* Uninvestigated hematuria or hematuria secondary to a malignant disease
* Clinically significant bladder outlet obstruction defined by clinical symptoms and investigator's opinion according to local standard of care (residual urine> 100mL of functional bladder capacity)
* Patients with marked cystocele or other clinically significant pelvic prolapse
* Treatment within 14 days preceding randomization, or expected to initiate treatment during the study with:

  * Any anticholinergic drugs other than a randomized trial drug
  * Any drug treatment for overactive bladder. Estrogen treatment started more than 2 months prior to inclusion is allowed
* On an unstable dosage of any drug with anticholinergic side effects, or expected to start such treatment during the study
* Receipt of any electrostimulation or bladder training within 14 days before randomization, or expected to start such treatment during the study
* An indwelling catheter or practicing intermittent self-catheterization
* Use of any investigational drug within 1 month prior to the start of the study
* Patients with chronic constipation or history of severe constipation
* Pregnant or nursing women
* Sexually active females of childbearing potential not using reliable contraception for at least 1 month prior to the start of the study and not agreeing to use such methods during the entire study period and for at least 1 month thereafter. Reliable contraceptive methods are defined as intrauterine devices (IUDs), combination type contraceptive pills, hormonal implants, double barrier method, injectable contraceptives and surgical procedures (tubal ligation or vasectomy)
* Patients who have bladder cancer or prostate cancer
* Treatment with potent CYP3A4 inhibitors, such as cyclosporine, vinblastine, macrolide antibiotics (e.g. erythromycin, clarithromycin, azithromycin) or antifungal agents (e.g. ketoconazole, itraconazole, micronazole)
* Patients who have neurological disease
* Patients who have psychological disease
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
change of micturition frequency on a 3-day voiding diary | after 12-week treatment

SECONDARY OUTCOMES:
change in patient's perception of bladder condition | after 12-week treatment
change in OAB symptom scores | after 12-week treatment
patient's satisfaction with the treatment | after 12-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Soo Choo, Professor, Principal Investigator — Asan Medical Center
Locations (6):
- South Korea (6):
  - Daegu
  - Daejeon
  - Inchon
  - Jeonnam
  - Pusan
  - Seoul

REFERENCES:
- [Derived] Han JY, Lee KS, Park WH, Park CH, Lee JG, Lee JZ, Kim DY, Na YG, Kwon DD, Choo MS. A comparative study on the efficacy of solifenacin succinate in patients with urinary frequency with or without urgency. PLoS One. 2014 Nov 17;9(11):e112063. doi: 10.1371/journal.pone.0112063. eCollection 2014. PMID 25401784